CLINICAL TRIAL: NCT01986595
Title: A Pilot Study on ALK Gene Mutations in Neuroblastoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201306008RINB
Record Dates: First submitted 2013-11-04; First posted 2013-11-18 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; anaplastic lymphoma kinase; cancer genetics; target therapy; RNA and genomic DNA extraction; complementary DNA(cDNA) preparation; Array-comparative genomic hybridization; Multiplex ligation-dependent probe amplification (MLPA); Sequencing of cDNA prepared from NB; Pyrosequencing; Quantitative real-time polymerase chain reaction(RT-PCR); Immunohistochemistry
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Biopsy tumor tissue(mail tumor or bone marrow) or Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Neuroblastoma (NB) originates from the sympathetic nervous system and is one of the most common cancers in infants and children. In our hospital, nearly 70% of patients are diagnosed with stage 4, metastatic disease with a poor prognosis, despite the use of multimodal therapy including chemotherapy, surgery, autologous stem cell transplantation, radiation therapy, and differentiation therapy. To improve the survival rate and patient care, our NB Study Group has devoted to the research on NB-specific molecular imaging, biomarkers, and target therapy. We have confirmed studies in cancer genetics by showing that N-myc gene (MYCN) amplification and segmental abnormalities on overall genomic profiling both have an adverse effect on treatment outcome. Therefore, there is an unmet need for the development of novel molecular target therapy in NB. Recently, the anaplastic lymphoma kinase (ALK) oncogene has been found to play an important role in the pathogenesis of NB, as well as serving as the driver mutations in approximately 10% of high-risk NB. The availability of ALK inhibitors also enables ALK as a treatment target in NB. In this proposal, we plan to utilize gene sequencing, array-comparative hybridization, and multiplex ligation-dependent probe amplification methods to evaluate the frequencies and characteristics of ALK mutations and amplifications in patients with NB. The gene and protein expression of ALK will also be evaluated by quantitative polymerase chain reaction(PCR) and immunohistochemistry, respectively, and compared with ALK genotype. The overall genomic pattern, clinical characteristics, histopathology, and treatment outcome of ALK-mutated NB patients will be analyzed. The results from this study may serve as the first report on ALK mutations of NB in Taiwan and will be used for the development of standardized genetic diagnosis protocols, as well as the design of future clinical trials targeting ALK.

DETAILED DESCRIPTION:
* purpose Despite the advance of modern multimodal therapy including surgery, chemotherapy, autologous stem cell transplantation, radiation therapy, and differentiation therapy, most children with NB are diagnosed with metastatic diseases and suffer from a dismal outcome. There is an unmet need for the development of novel target therapy in NB. Among all recently identified targets, ALK gene mutations have been found in approximately 10% of high-risk NB patients and are the treatment target of several promising agents that have already been tested in clinical trials, including crizotinib, which is to be available in Taiwan soon. This study aims to evaluate the prevalence of mutations and copy number aberrations of the ALK oncogene in prospective and previously treated NB patients' tumor sample (from surgical specimens) and germ-line (peripheral blood lymphocytes). The messenger ribonucleic acid(mRNA) and protein expression levels of ALK will also be analyzed. The results will be correlated with the clinical characteristics and pathological findings of this NB cohort.
* technique Prospective cases: Cryopreservation of tumor samples Retrospective cases: Archived tumor Sequencing: point mutation array-based comparative genomic hybridization(aCGH) & MLPA（multiplex ligation-dependent probe amplification）：analyze copy number alterations (CNAs) compare to clinical data
* expected results The results from this study may serve as the first report on ALK gene mutations of NB in Taiwan. We anticipate that 5-15% of NB tumors carry with common ALK mutations. Genome-wide CNAs profiling by aCGH can help us to categorize the genomic types of NB patients based on published guidelines, while the presence of ALK mutation or amplification may or may not be associated with subtypes with worse outcome. Some patients may have high ALK expression level without bearing common mutations on ALK gene locus, and we may identify novel mutation points in this patient cohort. Finally, we will probably find significant prognostic value of ALK gene mutation, which may be independent from other known risk factors, such as age, stage, MYCN amplification, and genomic pattern.

Based on these results, we are able to develop standardized protocol for diagnosing ALK mutations for Taiwanese NB patients. With the development of ALK genetic testing, a phase II clinical trial of an ALK inhibitor in high-risk NB patients with relapsed or refractory disease may subsequently be conducted and may improve the treatment outcome of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed by clinical criteria(one of below)

   Proved or maybe as Neuroblastoma by :
   1. pathological section
   2. Bone meta with 24 hrs urine Vanillylmandelic acid(VMA)or Homovanillic acid(HVA) elevated
   3. CT or MRI found tumor around adrenal gland or Neuroblastic tumor
2. Have tumor or blood samples to analyze ALK gene：

   1. will operation to remove tumor or biopsy, and will preserve tumor sample；or
   2. after operation and have tumor sample preserved；or
   3. after operation without tumor sample, but agree to take blood sample to analyze ALK mutation
3. Signed Inform Consent Form

Exclusion Criteria:

(1) After informed but still not consent

Max Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Neuroblastoma (NB) originates from the sympathetic nervous system and is one of the most common cancers in infants and children. In our hospital, nearly 70% of patients are diagnosed with stage 4, metastatic disease with a poor prognosis, despite the use of multimodal therapy including chemotherapy, surgery, autologous stem cell transplantation, radiation therapy, and differentiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
ALK gene mutations of NB in Taiwan | Baseline
  We anticipate that 5-15% of NB tumors carry with common ALK mutations. Genome-wide CNAs profiling by aCGH can help us to categorize the genomic types of NB patients based on published guidelines, while the presence of ALK mutation or amplification may or may not be associated with subtypes with worse outcome. Some patients may have high ALK expression level without bearing common mutations on ALK gene locus, and we may identify novel mutation points in this patient cohort. Finally, we will probably find significant prognostic value of ALK gene mutation, which may be independent from other known risk factors, such as age, stage, MYCN amplification, and genomic pattern.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Yao Lu, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Children Hospital, Taipei, Taiwan, Taiwan